CLINICAL TRIAL: NCT03658785
Title: Immunotherapy Using Precision T Cells Specific to Personalized Neo-antigen for the Treatment of Advanced Solid Tumor
Brief Title: Immunotherapy for the Treatment of Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wang Hui,MD, Vice Director of Deparment of Gynecology and Obstetrics, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018TNB-V01
Record Dates: First submitted 2018-09-03; First posted 2018-09-05 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Recurrence Tumor; Metastatic Cancer; Solid Tumor
Keywords: TIL; neo-antigen; Cyclophosphamide; Fludarabine
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TIL,IL-2,Cyclophosphamide,Fludarabine (Experimental): Biological: TIL On day 0, cells will be infused intravenously over 20 to 30 minutes (one to four days after the last dose of fludarabine).
  Drug: Aldesleukin 125,000 IU/kg IV/day (based on total body weight) beginning within 24 hours of cell infusion and continuing for up to 2 weeks) Drug: Cyclophosphamide On day -7 and day -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W over 1 hr.
  Drug: Fludarabine Days -5 to -1: Fludarabine 25 mg /m2/day IVPB daily over 30 minutes for 5 days.
  Interventions: Biological: TIL; Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: TIL — On day 0, cells will be infused intravenously over 20 to 30 minutes (one to four days after the last dose of fludarabine)
Drug: Aldesleukin — IL-2 125,000 IU/kg/day IV (based on total body weight) beginning within 24 hours of cell infusion and continuing for up to 2 weeks
  Other Names: IL-2
Drug: Cyclophosphamide — On day -7 and day -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W over 1 hr.
  Other Names: CTX
Drug: Fludarabine — Days -5 to -1: Fludarabine 25 mg /m2/day IVPB daily over 30 minutes for 5 days

SUMMARY:
The purpose of this study is to evaluate the safety, side effects and benefits of autologous tumor infiltrating lymphocytes (TIL) specific to personalized Neo-antigens in the treatment of patients with recurrent, metastatic and advanced solid tumors.

DETAILED DESCRIPTION:
Adoptive cell transfer therapy that utilizes an autologous TIL manufacturing progress is originally developed by the NCI for the treatment of patients with recurrent, metastatic cervical cancer and liver cancer. TILs specific to personalized neo-antigens will be expended in vitro and given back to the patients through vein. A total of 20 patients will be enrolled in the single-arm, open label, interventional study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients must meet ALL of the following criteria prior to enrollment in the study:

1. Must be ≥ 18 years of age at the time of consent.
2. Must have recurrent, metastatic, or persistent carcinoma that is not amenable to curative treatment with surgery and/or radiation therapy and for which no other therapies are expected to have significant benefit, in the opinion of the Investigator.
3. Must have at least 1 lesion that is resectable for TIL generation. The resected TIL generating lesion(s) should yield at least 1.5 cm in diameter post-resection of tumor tissue. Following resection for TIL generation, must have a remaining measurable target lesion as defined by RECIST v1.1.
4. Patients must have progressive disease while receiving or after the completion of the most recent prior treatment.
5. Any prior therapy directed at the malignant tumor must be discontinued at least 28 days prior to tumor resection. Radiation therapy may have been received up to 28 days prior to tumor resection for lesions not expected to be used for TIL generation or target lesions.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Patients must be seronegative for the human immunodeficiency virus (HIV).
8. Patients with positive serology for hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), or hepatitis C virus (anti-HCV) indicating acute or chronic infection may be enrolled if the viral load by polymerase chain reaction (PCR) is undetectable with/without active treatment.
9. Hematology:

   Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim;White blood cell (WBC) greater than or equal to 3000/mm(3);Platelet count greater than or equal too 100,000/mm(3);Hemoglobin greater than 8.0 g/dl.
10. Chemistry:

    Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to to 2.5 times the upper limit of normal. Serum creatinine less than or equal to to 1.6 mg/dl.Total bilirubin less that or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
11. Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.

Exclusion Criteria:

1. Patients who have received an organ allograft or prior cell transfer therapy.
2. Patients who are on a systemic steroid therapy > 10 mg of prednisone daily or other steroid equivalent.
3. Patients who currently have prior therapy-related toxicities greater than Grade 1 according to NCI-CTCAE v4.03; except for peripheral neuropathy, alopecia, or vitiligo prior to enrollment/resection.
4. Patients who have a contraindication to or history of hypersensitivity reaction to any component or excipients of the TIL therapy and the other study drugs.
5. Patients with active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory, or immune system.
6. Patients with symptomatic and/or untreated brain metastases (of any size and any number).
7. Patients who have any form of primary or acquired immunodeficiency syndrome, such as severe combined immunodeficiency disease or acquired immune deficiency syndrome (AIDS).
8. Patients who have a diagnosis of end-stage renal disorder requiring hemodialysis.
9. Patients who have a left ventricular ejection fraction (LVEF) < 45% or who are New York Heart Association (NYHA) Class 2 or higher.

   Patients who have a forced expiratory volume in 1 second (FEV1) of less than or equal to 60% of predicted normal.
10. Patients who have received a live or attenuated vaccine within 28 days of the NMA-LD regimen.
11. Patients whose cancer requires immediate treatment or who would otherwise suffer a disadvantage by participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Responce Rate [Time Frame: 24 months after cell infusion] | 24 months after cell infusion
  The Objective Responce Rate of patients received immunotherapy are accesed by the Response Criteria in Solid Tumors (RECIST) v1.0.

SECONDARY OUTCOMES:
Adverse Event | up to 24 months
  Aggregate of all adverse events, as well as their frequency and severity are accessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.03).
Disease Control Rate | up to 24 months
  Disease control rate (DCR) as measured by RECIST 1.1 criteria.
Duration of Response | up to 24 months
  Duration of response (DOR) as measured by RECIST 1.1 criteria .
Progression-Free Survival | up to 24 months
  PFS will be summarized using Kaplan-Meier estimates.
Overall Survival | up to 24 months
  The overall survival of all patients entering the study will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, MD, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stevanovic S, Draper LM, Langhan MM, Campbell TE, Kwong ML, Wunderlich JR, Dudley ME, Yang JC, Sherry RM, Kammula US, Restifo NP, Rosenberg SA, Hinrichs CS. Complete regression of metastatic cervical cancer after treatment with human papillomavirus-targeted tumor-infiltrating T cells. J Clin Oncol. 2015 May 10;33(14):1543-50. doi: 10.1200/JCO.2014.58.9093. Epub 2015 Mar 30. PMID 25823737
- [Background] Stevanovic S, Pasetto A, Helman SR, Gartner JJ, Prickett TD, Howie B, Robins HS, Robbins PF, Klebanoff CA, Rosenberg SA, Hinrichs CS. Landscape of immunogenic tumor antigens in successful immunotherapy of virally induced epithelial cancer. Science. 2017 Apr 14;356(6334):200-205. doi: 10.1126/science.aak9510. PMID 28408606
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Background] Zacharakis N, Chinnasamy H, Black M, Xu H, Lu YC, Zheng Z, Pasetto A, Langhan M, Shelton T, Prickett T, Gartner J, Jia L, Trebska-McGowan K, Somerville RP, Robbins PF, Rosenberg SA, Goff SL, Feldman SA. Immune recognition of somatic mutations leading to complete durable regression in metastatic breast cancer. Nat Med. 2018 Jun;24(6):724-730. doi: 10.1038/s41591-018-0040-8. Epub 2018 Jun 4. PMID 29867227